CLINICAL TRIAL: NCT01381913
Title: Feasibility Trial of Neoadjuvant Chemoradiotherapy in Patients With Locally Advanced Gastric Cancer Combined With Adjacent Tissue Invasion
Brief Title: Feasibility Trial of Neoadjuvant Chemoradiotherapy for Locally Advanced Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Kagawa University (Other)
Responsible Party: Tatsushi Inoue, Department of Gastroenterological Surgery, Faculty of Medicine, Kagawa University, Kagawa, Japan
Other Study IDs: NACRT-GC
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2005-10

CONDITIONS: Gastric Cancer; Chemoradiation
Keywords: Gastric cancer; Chemoradiotherapy; Adjacent tissue invasion; Feasibility trial
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Because locally far-advanced gastric cancer combined with adjacent tissue invasion has a poor prognosis, some phase 2 and 3 clinical trials of neoadjuvant chemotherapy (NAC) are performed in Japan. However, neoadjuvant chemoradiotherapy (NACRT) achieves superior local tumor control compared with NAC. This feasibility trial explored the feasibility and safety of neoadjuvant chemoradiotherapy (NACRT) in this type of gastric cancer.

DETAILED DESCRIPTION:
Since S-1 (combined drug of tegafur, 5-chloro-2,4-dihydroxypyridine and potassium oxonate) was approved in Japan in 1999 after a large-scale clinical trial, adjuvant chemotherapy with S-1 has been the standard treatment for stage II/III gastric cancer. However, for far-advanced gastric cancer, various adjuvant chemotherapies, including S-1, have not achieved satisfactory results. Therefore, Japan Clinical Oncology Group (JCOG) is currently performing phase 2 and 3 clinical trials of neoadjuvant chemotherapy (NAC) for locally far-advanced gastric cancer. However, previous studies of NAC have reported a pathological response rate of 15-50% for the main lesion, indicating no significant effect on local tumor control.

On the other hand, other studies have reported that anticancer drugs, including S-1, have a radiosensitizing effect, and that neoadjuvant chemoradiotherapy (NACRT) achieves superior local tumor control compared with NAC. Therefore, we conducted a feasibility trial of NACRT with S-1 for locally far-advanced gastric cancer combined with adjacent tissue invasion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric adenocarcinoma
* Tumor invasion of adjacent structures (T4) and/or tumors with bulky nodal metastases
* No metastases outside of Group 2 lymph nodes
* Neither peritoneal metastasis nor liver metastasis
* No other distant metastasis
* An Eastern cooperative oncology group performance status of between 0 and 2
* No prior radiation therapy
* Sufficient organ function

Exclusion Criteria:

* A synchronous or previously active malignancy
* Insufficient oral intake
* A history of severe allergy
* Watery diarrhea
* Severe co-morbidities
* Requiring therapy for pericardial effusion or pleural effusion
* Contraindications to S-1 or radiotherapy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Histologically proven gastric adenocarcinoma
  * Tumor invasion of adjacent structures (T4) and/or tumors with bulky nodal metastases
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Yachida, M. D. Ph. D., Study Director — Department of Gastroenterological Surgery, Faculty of Medicine, Kagawa University, Kagawa, Japan; Yasuyuki Suzuki, M. D. Ph. D., Principal Investigator — Department of Gastroenterological Surgery, Faculty of Medicine, Kagawa University, Kagawa, Japan
Locations (1):
- Department of Gastroenterological Surgery, Faculty of Medicine, Kagawa University, Kita, Kagawa-ken, Japan